CLINICAL TRIAL: NCT05670847
Title: Efficacy of Ketone Esters for Children With Drug Resistant Epilepsy
Brief Title: Exogenous Ketone Esters for Drug Resistant Epilepsy
Acronym: EKEDRE
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Elsayed Abdelkreem, Lecturer of Pediatrics, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-22-12-45
Record Dates: First submitted 2022-12-18; First posted 2023-01-04 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Drug Resistant Epilepsy
Keywords: Drug resistant epilepsy; Exogenous ketone esters; Children
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Intervention Model Description: Eligible children will be randomized into two equal-sized groups. Study group: will receive exogenous ketone esters plus standard of care. Control group: will receive only standard of care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Children receiving exogenous ketone esters + standard of care
  Interventions: Drug: Exogenous ketone ester
- Control group (No Intervention): Children receiving only standard of care

INTERVENTIONS:
Drug: Exogenous ketone ester — 500 mg/kg orally three times daily (with at least 4 hours between each dose) for 28 days
  Arms: Study group

SUMMARY:
This study aims to investigate the efficacy of add-on exogenous ketone esters for treating children with drug-resistant epilepsy

DETAILED DESCRIPTION:
Epilepsy is a common neurological disorder among children with significant neurobiological, cognitive, psychological, and social consequences. Seizures can usually be controlled by anti-seizure medications (ASMs) in up to two-thirds of children with epilepsy. However, this leaves a significant part of epileptic children whose seizures are not controlled by pharmacotherapy. Currently, available alternatives for drug-resistant epilepsy (DRE) include surgery, vagus nerve stimulation, and ketogenic diet (KD).

KD has been classically used for treating children with DRE. However, KD requires strict dietary restriction, which may not be applicable or acceptable for many patients, and is associated with several adverse effects, commonly including gastrointestinal (e.g., constipation, nausea, vomiting), cardiovascular (e.g., dyslipidemia), renal/genitourinary (e.g., renal calculi), and growth problems. Exogenous ketone esters (EKE) could be a more convenient and superior alternative to KD for children with DRE.

ELIGIBILITY:
Inclusion Criteria:

* Drug-resistant epilepsy
* Seizure frequency ≥ 7 per week

Exclusion Criteria:

* Failure to obtain informed consent
* Recent intake of exogenous ketones, ketogenic diet, or any dietary restrictions/modifications
* Severe disease conditions, including hepatic, renal, respiratory, cardiac, gastrointestinal, endocrinal, and immune systems
* Hypo-/hyperglycemia
* Metabolic acidosis
* Ketosis (βHB > 2 mmol/L)
* GIT disorders, including gastritis/peptic ulcer, diarrhea/constipation, and irritable bowel disease
* Malnutrition/obesity
* Limitations to oral feeding (e.g., severe gastroesophageal reflux)
* Inborn errors of metabolism
* Chromosomal disorders
* Surgically-remediable epilepsy
* Allergies or any other contraindication to ketone supplements
* Inapplicable recording of seizures
* Incompliance to anti-seizure medications and/or irregular follow-up
* Recent propofol therapy
* Intake of carbonic-anhydrase inhibitors

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
≥ 50% reduction in seizure frequency | From 28-days observation (baseline) phase to 28-days intervention phase
  Proportion of patients achieving ≥ 50% reduction in seizure frequency

SECONDARY OUTCOMES:
Proportion of incompliance to exogenous ketone ester therapy | 28-days intervention phase
  Proportion of doses of exogenous ketone esters which were not administered by patients (as recorded by parents of included children)
Proportion of incompliance to anti-seizure medications (ASMs) | From 28-days observation (baseline) phase to 28-days intervention phase
  Proportion of doses of anti-seizure medications (ASMs) which were not administered by children (as recorded by parents of included children)
Change in seizure severity assessed by National Hospital Seizure Severity Scale (NHS3) | From 28-days observation (baseline) phase to 28-days intervention phase
  Change in seizure severity assessed by National Hospital Seizure Severity Scale (NHS3)
Change in seizure frequency | From 28-days observation (baseline) phase to 28-days intervention phase
  Change in the number of seizures (as recorded by parents of included children)
Change in frequency of status epilepticus | From 28-days observation (baseline) phase to 28-days intervention phase
  Change in the number of episodes of status epilepticus (evaluated from patient's medical records)
Change in occurrence of possible adverse effects | From 28-days observation (baseline) phase to 28-days intervention phase
  Change in occurrence of possible adverse effects
Change in cognitive domains | From 28-days observation (baseline) phase to 28-days intervention phase
  Change in attention, alertness, and memmory, each rated by parents of included children at the end of 28-days intervention phase as no change, improvement, or regression in comparison with the preceding 28-days observation phase
Change in blood βHB | From baseline to 30 minutes, 1 hour, 2 hours, 4 hours, 2 days, 4 days, 7 days, 14 days, and 28 days study timepoints
  Change in blood level of beta-hydroxybutyrate
Change in blood glucose | From baseline to 30 minutes, 1 hour, 2 hours, 4 hours, 2 days, 4 days, 7 days, 14 days, and 28 days study timepoints
  Change in blood level of glucose
Change in blood pH | From baseline to 30 minutes, 1 hour, 2 hours, 4 hours, 2 days, 4 days, 7 days, 14 days, and 28 days study timepoints
  Change in blood level of pH
Change in EEG score | From baseline to 28 days study timepoint
  Change in EEG score according to the scale developed by Walker & Said (2014), which includes items related to encephalopathy, interictal epileptic discharge, and seizure presence

OTHER OUTCOMES:
Change in blood lactate level | From baseline to 30 minutes, 1 hour, 2 hours, 4 hours, 2 days, 4 days, 7 days, 14 days, and 28 days study timepoints
  Change in blood level of lactate
Change in blood bicarbonate level | From baseline to 30 minutes, 1 hour, 2 hours, 4 hours, 2 days, 4 days, 7 days, 14 days, and 28 days study timepoints
  Change in blood level of bicarbonate
Change in serum sodium level | From baseline to 30 minutes, 1 hour, 2 hours, 4 hours, 2 days, 4 days, 7 days, 14 days, and 28 days study timepoints
  Change in serum sodium level
Change in serum potassium level | From baseline to 30 minutes, 1 hour, 2 hours, 4 hours, 2 days, 4 days, 7 days, 14 days, and 28 days study timepoints
  Change in serum potassium level
Change in hematological counts | From baseline to 28 days study timepoint
  Change in hematological counts
Change in blood triglycerides level | From baseline to 28 days study timepoint
  Change in blood triglycerides level
Change in blood free fatty acids level | From baseline to 28 days study timepoint
  Change in blood free fatty acids level
Change in blood cholesterol level | From baseline to 28 days study timepoint
  Change in blood cholesterol level
Change in HbA1c | From baseline to 28 days study timepoint
  Change in hbA1c
Change in blood alanine transaminase level | From baseline to 28 days study timepoint
  Change in blood level of alanine transaminase enzyme (ALT)
Change in serum creatinine level | From baseline to 28 days study timepoint
  Change in serum level of creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Abdelrahim A Sadek, MD, PhD, Study Chair — Sohag University
Locations (1):
- Department of Pediatrics at Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Unidentified individual participant data (IPD) underlying study results will be available upon reasonable request
Supporting Information: Study Protocol, SAP
Time Frame: Unidentified individual participant data (IPD) underlying study results will be available upon reasonable request 6-months after publication

REFERENCES:
- [Background] Carson RP, Herber DL, Pan Z, Phibbs F, Key AP, Gouelle A, Ergish P, Armour EA, Patel S, Duis J. Nutritional Formulation for Patients with Angelman Syndrome: A Randomized, Double-Blind, Placebo-Controlled Study of Exogenous Ketones. J Nutr. 2021 Dec 3;151(12):3628-3636. doi: 10.1093/jn/nxab284. PMID 34510212
- [Background] Clarke K, Tchabanenko K, Pawlosky R, Carter E, Todd King M, Musa-Veloso K, Ho M, Roberts A, Robertson J, Vanitallie TB, Veech RL. Kinetics, safety and tolerability of (R)-3-hydroxybutyl (R)-3-hydroxybutyrate in healthy adult subjects. Regul Toxicol Pharmacol. 2012 Aug;63(3):401-8. doi: 10.1016/j.yrtph.2012.04.008. Epub 2012 May 3. PMID 22561291
- [Background] Stubbs BJ, Cox PJ, Evans RD, Santer P, Miller JJ, Faull OK, Magor-Elliott S, Hiyama S, Stirling M, Clarke K. On the Metabolism of Exogenous Ketones in Humans. Front Physiol. 2017 Oct 30;8:848. doi: 10.3389/fphys.2017.00848. eCollection 2017. PMID 29163194
- [Background] Cox PJ, Kirk T, Ashmore T, Willerton K, Evans R, Smith A, Murray AJ, Stubbs B, West J, McLure SW, King MT, Dodd MS, Holloway C, Neubauer S, Drawer S, Veech RL, Griffin JL, Clarke K. Nutritional Ketosis Alters Fuel Preference and Thereby Endurance Performance in Athletes. Cell Metab. 2016 Aug 9;24(2):256-68. doi: 10.1016/j.cmet.2016.07.010. Epub 2016 Jul 27. PMID 27475046
- [Background] Gilbert DL, Pyzik PL, Freeman JM. The ketogenic diet: seizure control correlates better with serum beta-hydroxybutyrate than with urine ketones. J Child Neurol. 2000 Dec;15(12):787-90. doi: 10.1177/088307380001501203. PMID 11198492
- [Background] Kwan P, Arzimanoglou A, Berg AT, Brodie MJ, Allen Hauser W, Mathern G, Moshe SL, Perucca E, Wiebe S, French J. Definition of drug resistant epilepsy: consensus proposal by the ad hoc Task Force of the ILAE Commission on Therapeutic Strategies. Epilepsia. 2010 Jun;51(6):1069-77. doi: 10.1111/j.1528-1167.2009.02397.x. Epub 2009 Nov 3. PMID 19889013
- [Background] Scheffer IE, Berkovic S, Capovilla G, Connolly MB, French J, Guilhoto L, Hirsch E, Jain S, Mathern GW, Moshe SL, Nordli DR, Perucca E, Tomson T, Wiebe S, Zhang YH, Zuberi SM. ILAE classification of the epilepsies: Position paper of the ILAE Commission for Classification and Terminology. Epilepsia. 2017 Apr;58(4):512-521. doi: 10.1111/epi.13709. Epub 2017 Mar 8. PMID 28276062
- [Background] Walker I, Said RR. Predictors of Ketogenic Diet Efficacy in Children Based on the Electroencephalogram (EEG). J Child Neurol. 2015 Sep;30(10):1270-4. doi: 10.1177/0883073814556888. Epub 2014 Nov 20. PMID 25414234